CLINICAL TRIAL: NCT05348304
Title: Hypoglycemic Effects of a Dietary Supplement That Combines the Properties of Myo-inositol and D-chiro-inositol With Gymnema Silvestre, Alpha-lactalbumin and Zinc.
Brief Title: Hypoglycemic Effects of a Dietary Supplement With Inositols, Gymnema Silvestre, Alpha-lactalbumin and Zinc.
Acronym: EUDIA_22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EUDIA_22
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-06

CONDITIONS: Metabolism Disorder
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Hypocaloric diet
- EUDIAMET (Experimental): Hypocaloric diet plus a supplementation with myo-inositol and D-chiro-inositol in the 40:1 ratio, Gymnema sylvestre, alpha-lactalbumin and zinc
  Interventions: Dietary Supplement: EUDIAMET

INTERVENTIONS:
Dietary Supplement: EUDIAMET — A combination of myo-inositol and D-chiro-inositol in the 40:1 ratio, Gymnema sylvestre, alpha-lactalbumin and zinc
  Arms: EUDIAMET

SUMMARY:
This study is aimed at evaluating the hypoglycemic effects of a dietary supplement that associates the properties of two inositols (myo-inositol and D-chiro-inositol) in the ratio 40:1 to Gymnema sylvestre, alpha-lactalbumin and zinc.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 35
* Basal Glycemia between 100 and 125 mg/dl

Exclusion Criteria:

* Diabetes diagnosis
* Use of food supplements containing inositols, gymnema, alpha-lactalbumin and zinc
* Intolerance to inositols, gymnema, alpha-lactalbumin and zinc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Insulinemia | Three time points: change in insulin levels from the baseline to three and six months
  Reduction of systemic insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Basciani, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No